CLINICAL TRIAL: NCT01970111
Title: An Extension Study of KPS-0373 in Patients With Spinocerebellar Degeneration (SCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KPS1302
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Spinocerebellar Degeneration
Keywords: Spinocerebellar degeneration (SCD); Thyrotropin-Releasing Hormone (TRH); Spinocerebellar Ataxia (SCA); Cortical Cerebellar Atrophy (CCA)
MeSH Terms: conditions — Spinocerebellar Degenerations; Spinocerebellar Ataxias

ARMS (1):
- KPS-0373 (Experimental)
  Interventions: Drug: KPS-0373, High dose; Drug: KPS-0373, Low dose

INTERVENTIONS:
Drug: KPS-0373, High dose
Drug: KPS-0373, Low dose

SUMMARY:
The purpose of this study is to evaluate the long-term safety, efficacy, and pharmacokinetics of KPS-0373 in SCD patients.

ELIGIBILITY:
Inclusion Criteria:

* Japanese SCD patients with mild to moderate ataxia (Completion of the KPS1301 study)

Exclusion Criteria:

* Less than 75% of compliance in KPS1301 study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
SARA (Scale for the Assessment and Rating of Ataxia) | 52 weeks

SECONDARY OUTCOMES:
SF-8 (QOL) | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo and Other Japanese Cities, Japan